CLINICAL TRIAL: NCT06166186
Title: Effect of Intraoperative Music on Inflammatory Response in Adult Living Donor Hepatectomy.
Brief Title: Effect of Intraoperative Music on Inflammatory Response in Donor Hepatectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istinye University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: anestezi3
Record Dates: First submitted 2023-11-14; First posted 2023-12-12 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2023-10

CONDITIONS: Transplantation; Hepatectomy; Music; Stress Response
MeSH Terms: conditions — Fractures, Stress | interventions — Music Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music Group (Active Comparator): Music will be delivered via headphones intraoperatively. Blood samples will be collected as per the protocol.
  Interventions: Other: music
- Control Group (Active Comparator): Headphones will be applied but no music will be played intraoperatively. Blood samples will be collected as per the protocol.
  Interventions: Other: no music

INTERVENTIONS:
Other: music — A music with a standard volume will be delivered to the patients via headphones from the beginning of anesthesia induction to extubation.
  Arms: Music Group
Other: no music — Headphones will be applied to the patients but no music will be played from the beginning of anesthesia induction to extubation.
  Arms: Control Group

SUMMARY:
It has been reported that non-pharmacological methods can be used as an alternative in addition to pharmacological methods to reduce pain, anxiety, stress and inflammatory response that begins with the surgical incision in the intraoperative period and continues throughout the operation. It has been reported that music can be used as an alternative non-pharmacological method to reduce pain and anxiety in the perioperative period, as well as surgical stress and the related stress response.

The aim of this study is to test the hypothesis that music used as a non-pharmacological method in the intraoperative period can reduce inflammatory response in living donor hepatectomy.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing donor hepatectomy
* American Society of Anesthesiologists class 1 to 2
* Ability to consent

Exclusion Criteria:

* American Society of Anesthesiologists greater than 2
* Documented or known sensitivity to any drug to be used in the study.
* Patient with immunosuppressant/ cytotoxic/ steroid therapy.
* not understand the aim and objectives of the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2023-05-22 (Actual); Primary Completion 2024-07-12 (Actual); Study Completion 2024-09-09 (Actual)

PRIMARY OUTCOMES:
Differences in Interleukin-6 (IL-6) | 4 hours
  Serum levels of IL-6 will be measured preoperatively and postoperatively.

SECONDARY OUTCOMES:
Difference in tumor necrosis factor alpha (TNF-alfa) | 4 hours
  Serum levels of TNF-alpha will be measured preoperatively and postoperatively.
Difference between serum levels of total antioxidant capacity (TAC) at preoperative and postoperative period. | 4 hours
  Blood samples will be collected preoperatively and postoperatively to measure serum levels of TAC. Blood samples will be stored in medical refrigerator and analysis for serum levels of TAC will be done after collection of all samples.
Difference between serum levels of total oxidant capacity (TOC) at preoperative and postoperative period. | 4 hours
  Blood samples will be collected preoperatively and postoperatively to measure serum levels of TOC. Blood samples will be stored in medical refrigerator and analysis for serum levels of TOC will be done after collection of all samples.
Difference in c-reactive protein (CRP) | 24 hours
  Serum levels of CRP will be measured preoperatively and postoperatively.
Difference in alanine aminotransferase (ALT) | 24 hours
  Serum levels of ALT will be measured preoperatively and postoperatively.
Difference in aspartate aminotransferase (AST) | 24 hours
  Serum levels of AST will be measured preoperatively and postoperatively.
Difference in creatinine | 24 hours
  Serum levels of creatinine will be measured preoperatively and postoperatively.
Differences in preoperative State-Trait Anxiety Inventory scores | 20 minutes
  assessed 1 day before surgery. The total score on the scale ranges from 20 to 80 points and a higher score represents greater anxiety.
Differences in postoperative State-Trait Anxiety Inventory scores | 20 minutes
  assessed 1st day after surgery. The total score on the scale ranges from 20 to 80 points and a higher score represents greater anxiety.
Differences in pain scores | 24 hours
  Assessed 1st, 6th, 12th and 24th hour postoperatively. (from 0 (no pain) to 10 (maximal possible pain))

CONTACTS AND LOCATIONS:
Overall Officials: Beyza Zeynep Kocabicak, Principal Investigator — Istinye University; Ali Sait Kavakli, M.D., Principal Investigator — Istinye University; Taylan Sahin, M.D., Principal Investigator — İstinye University
Locations (1):
- Istinye University Hospital, Istanbul, Turkey (Türkiye)